CLINICAL TRIAL: NCT06987838
Title: Effect of Virtual Reality on Prostaglandin Levels in Adolescent Females With Primary Dysmenorrhea: A Randomized Controlled Trial
Brief Title: Effect of Virtual Reality on Prostaglandin Levels in Adolescent Females With Primary Dysmenorrhea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha National University (Other)
Responsible Party: Principal Investigator, Sally Mohamed Saeed, Principal Investigator, Benha National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005600
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Primary Dysmenorrhea
MeSH Terms: interventions — Drug Therapy; Ibuprofen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacological treatment (Other): It will consist of 25 girls, who will receive pharmacological treatment in the form of ibuprofen 400 mg, three times per day, during the first 2 days of menstruation, for 3 menstrual cycles.
  Interventions: Drug: Pharmacological treatment
- Virtual reality + Pharmacological treatment (Experimental): It will consist of 25 girls, who will receive the same pharmacological treatment in addition to virtual reality during the first 2 days of menstruation, for 3 menstrual cycles.
  Interventions: Drug: Pharmacological treatment; Other: Virtual reality

INTERVENTIONS:
Drug: Pharmacological treatment — All participants in the two groups will receive pharmacological treatment in the form of ibuprofen 400 mg, three times per day, during the first 2 days of menstruation, for 3 menstrual cycles.
  Other Names: Ibuprofen (400 mg)
Other: Virtual reality — The experimental group will receive virtual reality during the first 2 days of menstruation, for 3 menstrual cycles.
  Arms: Virtual reality + Pharmacological treatment

SUMMARY:
This study will be conducted to study the effect of virtual reality therapy on prostaglandin levels in adolescent females with primary dysmenorrhea.

DETAILED DESCRIPTION:
Primary dysmenorrhea is thought to be caused by excessive levels of prostaglandins, which are hormones that stimulate the uterus to contract during menstruation and childbirth, Treatment must be tailored to individual patient symptoms. Pharmacologic management with non-steroidal anti-inflammatory medications and/or combined hormonal contraceptives is most common. Heat therapy, exercise, vitamins and dietary supplements have limited evidence and can be offered for patients seeking non-pharmacologic adjunctive or alternative options. Greater awareness for both health-care providers and patients allow for early intervention to reduce impact on quality of life and life course potential. The significance of this study to assess the effect of virtual reality therapy on primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Age 17- 21 years old.
* The body mass index (BMI) < 30 kg/m2.
* Unmarried females.
* Females with dysmenorrhea pain.
* Females with regular menstrual cycles.
* Females with normal gynecology.

Exclusion Criteria:

* Have a pathological disease related to reproduction.
* Students who use analgesic drugs for 3 months/3 menstrual cycles.
* Students with menstrual pain secondary to diagnosed organic or inflammatory causes.

Ages: 17 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-25 (Estimated); Primary Completion 2025-08-25 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 12 weeks
  Participants in both groups will complete the visual analogue scale (VAS) before the start of treatment and after 3 menstrual cycles of treatment. The VAS is a 10 cm horizontal line on which the participants' pain intensity is represented by a point between the extremes of "no pain at all "and "worst pain imaginable". Each girl will be asked to mark a point on the line between the extreme that was related to her pain intensity. Then, the distance will be measured each time from the left end of the line to the marked point to obtain the VAS score for pain intensity of dysmenorrhea.
Assessment of Prostaglandin Levels | 12 weeks
  Blood samples will be collected from each girl in both groups to measure the levels of plasma PGF2α before the start of treatment and after 3 menstrual cycles of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sally Mohamed Saeed, PhD, Principal Investigator — Lecturer, Benha National University; Malak Adel El Mahdy, PhD, Principal Investigator — Lecturer, Al Hayah University; Sarah Abdullah Mohamed Elsamahy, PhD, PhD, Principal Investigator — Lecturer, Misr University for Science and Technology; Samah Mahmoud Ahmed sheha, PhD, Principal Investigator — Lecturer, Misr University for Science and Technology; Naglaa fathey moustafa, PhD, Principal Investigator — Lecturer, Al Hayah University
Locations (1):
- Misr University for Science and Technology, Giza, Egypt